CLINICAL TRIAL: NCT01026454
Title: A Randomized, Open-label, Crossover Trial of the Effect of High-dose Daily HSV-2 Suppressive Therapy on Plasma HIV-1 Levels Among HIV-1/HSV-2 Co-infected Persons
Brief Title: Valacyclovir vs. Acyclovir as HSV-2 Suppressive Therapy: Effect on Plasma HIV-1 Levels Among HIV-1/HSV-2 Co-infected Persons
Acronym: ACV-VAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Connie Celum, US Principal Investigator, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 37162-A
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: HSV Infection; HIV Infection
Keywords: HSV; HIV
MeSH Terms: conditions — Herpes Simplex; HIV Infections | interventions — Acyclovir; Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acyclovir (Active Comparator): acyclovir 400 mg orally twice daily
  Interventions: Drug: acyclovir
- valacyclovir (Active Comparator): valacyclovir 1.5 g orally twice daily
  Interventions: Drug: valacyclovir

INTERVENTIONS:
Drug: acyclovir — acyclovir 400 mg orally, twice daily for 12 weeks
  Arms: acyclovir
Drug: valacyclovir — valacyclovir 1.5 g orally, twice daily, for 12 weeks
  Arms: valacyclovir

SUMMARY:
The purpose of this study is to determine whether treating HSV-2 with either valacyclovir or acyclovir is more effective in suppressing HIV-1 virus levels in people co-infected with HIV-1 and HSV-2.

DETAILED DESCRIPTION:
Sexual transmission is responsible for the vast majority of HIV-1 infections among adults worldwide. In sub-Saharan Africa, the region hardest hit by the HIV-1 epidemic, HSV-2 prevalences of 30-50% have been seen in the general population with prevalence up to 90% in infected with HIV-1. HSV-2 is common in those with, or at risk for, HIV-1 infection, and HSV-2 reactivation increases HIV-1 acquisition and infectiousness. Recent studies have shown that suppression of HSV-2 has a sustained effect on lowering HIV-1 levels in blood plasma. New data have raised the question whether higher doses of HSV-2 suppressive therapy might be more effective at suppressing HIV-1 levels. Acyclovir and valacyclovir, chosen for use in this study, are safe and effective treatments for decreasing the frequency of HSV-2 reactivation and shedding. The standard dose of acyclovir is 400 mg twice a day. Valacyclovir, a drug that converts to acyclovir after absorption, delivers higher concentrations of acyclovir. 1.5 grams of valacyclovir, will be used to provide a higher dose of acyclovir, and will be compared with the standard dose of 400 mg twice a day of acyclovir.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive
* Not on HIV-1 antiretroviral therapy nor planning to initiate antiretroviral therapy during the study period
* CD4 cell count >250 cell/µL
* Not otherwise eligible for antiretroviral therapy according to Uganda national guidelines
* Detectable HIV-1 plasma viral load
* HSV-2 seropositive
* Not intending to move out of the area for the duration of study participation.
* Able to participate in the study at the Partners in Prevention site in Thika, Kenya

Exclusion Criteria:

* Known history of adverse reaction to acyclovir, valacyclovir, or famciclovir.
* Planned use of acyclovir, valacyclovir, or famciclovir
* Use of ganciclovir, foscarnet, or cidofovir
* Known medical history of seizures
* Serum creatinine >1.5 mg/dL
* AST or ALT >3 times upper limit of normal
* Hematocrit <30 %
* Absolute neutrophil count <1000
* Platelet count <75,000
* History of thrombotic microangiopathy
* Any other condition which, in the opinion of the principal investigator, may compromise the ability to follow study procedures and complete the study
* Participation in another HIV therapeutics trial
* For women, pregnancy as confirmed by a urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Thika Partners in Prevention, Thika, Kenya

REFERENCES:
- [Background] Brown EL, Wald A, Hughes JP, Morrow RA, Krantz E, Mayer K, Buchbinder S, Koblin B, Celum C. High risk of human immunodeficiency virus in men who have sex with men with herpes simplex virus type 2 in the EXPLORE study. Am J Epidemiol. 2006 Oct 15;164(8):733-41. doi: 10.1093/aje/kwj270. Epub 2006 Aug 8. PMID 16896053
- [Background] Freeman EE, Weiss HA, Glynn JR, Cross PL, Whitworth JA, Hayes RJ. Herpes simplex virus 2 infection increases HIV acquisition in men and women: systematic review and meta-analysis of longitudinal studies. AIDS. 2006 Jan 2;20(1):73-83. doi: 10.1097/01.aids.0000198081.09337.a7. PMID 16327322
- [Background] Schacker T, Zeh J, Hu H, Shaughnessy M, Corey L. Changes in plasma human immunodeficiency virus type 1 RNA associated with herpes simplex virus reactivation and suppression. J Infect Dis. 2002 Dec 15;186(12):1718-25. doi: 10.1086/345771. Epub 2002 Nov 22. PMID 12447756
- [Derived] Mugwanya K, Baeten JM, Mugo NR, Irungu E, Ngure K, Celum C. High-dose valacyclovir HSV-2 suppression results in greater reduction in plasma HIV-1 levels compared with standard dose acyclovir among HIV-1/HSV-2 coinfected persons: a randomized, crossover trial. J Infect Dis. 2011 Dec 15;204(12):1912-7. doi: 10.1093/infdis/jir649. Epub 2011 Oct 12. PMID 21998479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HSV-2/HIV-1 dually-infected participants were recruited between March and November 2010 from Thika, Kenya.
Pre-assignment Details: 66 participants screened; 34 excluded (33 did not meet inclusion criteria, 1 declined study participation); 32 enrolled
Groups:
- Acyclovir Then Valacyclovir: Acyclovir 400 mg orally twice daily (12 weeks), Washout (2 weeks), Valacyclovir 1.5 g orally twice daily (12 weeks)
- Valacyclovir Then Acyclovir: Valacyclovir 1.5 g orally twice daily (12 weeks), Washout (2 weeks), Acyclovir 400 mg orally twice daily (12 weeks)
Period: First Intervention
Arm/Group | Acyclovir Then Valacyclovir | Valacyclovir Then Acyclovir
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: Washout
Arm/Group | Acyclovir Then Valacyclovir | Valacyclovir Then Acyclovir
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Acyclovir Then Valacyclovir | Valacyclovir Then Acyclovir
Started | 17 | 14
Completed | 16 | 13
Not Completed | 1 | 1
Not completed — Pregnancy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Acyclovir Then Valacyclovir: acyclovir 400 mg orally twice daily for 12 weeks, 2 week washout, then valacyclovir 1.5 g orally twice daily for 12 weeks
- Valacyclovir Then Acyclovir: valacyclovir 1.5 g orally twice daily for 12 weeks, 2 week washout, then acyclovir 400 mg orally twice daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Acyclovir Then Valacyclovir | Valacyclovir Then Acyclovir | Total
Number analyzed (Participants) | 18 | 14 | 32
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 14 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Kenya | 18 | 14 | 32
Plasma HIV-1 RNA Level at Enrollment [Mean (Standard Deviation); unit: log10 copies/mL] | 4.05 (0.72) | 4.08 (0.85) | 4.07 (0.75)

OUTCOME MEASURES:

1. Primary Outcome: Mean Level of HIV-1 RNA in Plasma of Participants While on Acyclovir or Valacyclovir.
Description: Mean level of HIV-1 RNA in plasma of participants while on 400 mg twice daily of acyclovir versus while on 1.5 g twice daily of valacyclovir.
Time Frame: Weekly for 12 weeks per intervention
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Groups:
- Acyclovir: acyclovir 400 mg twice daily 400 mg either in first intervention period or second
- Valacyclovir: valacyclovir 1.5 g twice daily either in first intervention period or second
Arm/Group | Acyclovir | Valacyclovir
Number analyzed (Participants) | 32 | 31
log10 copies/mL | 3.56 [3.26 to 3.85] | 2.94 [2.65 to 3.24]

2. Secondary Outcome: Safety of Valacyclovir 1.5 Gram Orally Twice Daily in HIV-1 Seropositive Persons.
Time Frame: 28 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Acyclovir | Valacyclovir
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No